CLINICAL TRIAL: NCT05187910
Title: Correlation Between Montreal Cognitive Assessment and Voice Therapy Outcomes in the Aging Treatment- Seeking Population
Acronym: MoCA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Emory University (Other); New York University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 20-29913
Record Dates: First submitted 2021-11-04; First posted 2022-01-12 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: Cognitive Impairment; Voice Disorders; Voicebox Disorders; Cognitive Decline; Swallowing Disorder
Keywords: voice therapy; cough therapy; swallowing therapy
MeSH Terms: conditions — Cognitive Dysfunction; Voice Disorders; Deglutition Disorders | interventions — Speech Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Patients with Voice Disorders (Active Comparator): This is typically diagnosed by MDs in conjunction with Speech Language Pathologists (SLPs).
  Interventions: Behavioral: Speech Therapy
- Patients with Swallowing Disorders (Active Comparator): This is typically diagnosed by MDs in conjunction with Speech Language Pathologists (SLPs).
  Interventions: Behavioral: Swallowing Therapy
- Patients with Upper Airway Disorders (Active Comparator): This is typically diagnosed by MDs in conjunction with Speech Language Pathologists (SLPs).
  Interventions: Behavioral: Upper Airway Therapy

INTERVENTIONS:
Behavioral: Speech Therapy — Training with a Speech Language Pathologists for voice disorders. This is typically done with an initial visit done jointly with an MD physician. Then there are 4 subsequent therapy visits in addition to home practice exercises. Finally there will be another joint post-treatment evaluation to determine progress and next steps.
  Arms: Patients with Voice Disorders
Behavioral: Swallowing Therapy — Training with a Speech Language Pathologists for swallowing disorders. This is typically done with an initial visit done jointly with an MD physician. Then there are 4 subsequent therapy visits in addition to home practice exercises. Finally there will be another joint post-treatment evaluation to determine progress and next steps.
  Arms: Patients with Swallowing Disorders
Behavioral: Upper Airway Therapy — Training with a Speech Language Pathologists for upper airway disorders. This is typically done with an initial visit done jointly with an MD physician. Then there are 4 subsequent therapy visits in addition to home practice exercises. Finally there will be another joint post-treatment evaluation to determine progress and next steps.
  Arms: Patients with Upper Airway Disorders

SUMMARY:
This study will investigate if the performance on the Montreal Cognitive Assessment (MoCA) is associated or predictive of the outcomes in voice, swallowing or upper airway therapy in the older laryngology treatment seeking patients. The relationship between the scores of MoCA and parameters in therapy will be analyzed. The outcomes of this study could potentially impact how investigators determine candidacy for therapy and develop patient treatment plans to meet their needs. This is a collaborative study with Emory Voice Center and the NYU Voice Center.

ELIGIBILITY:
Inclusion Criteria:

* 60 years or older with voice/swallowing/upper airway complaints
* Multidisciplinary assessment by fellowship-trained laryngologist and voice/swallow/upper airway specialized speech-language pathologist
* Voice, Swallowing and/or Upper airway disorder diagnosis
* Candidate for voice, swallowing or upper airway therapy following interdisciplinary assessment.
* State willingness to participate in the study protocol

Exclusion Criteria:

* Under the age of 60 years old
* Previously diagnosed dementia
* Central neurological disorder
* Active psychotic disorder
* Recurrent or active major depressive disorder (PHQ-9 of 10 or greater)
* Patient not able to attempt the MoCA because of a severe hearing or visual impairment
* Patients who do not speak or understand English
* Tested with MoCA in the last month

Ages: 60 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
Change in Voice Handicap Index-10 Score Following Therapy | Recorded at initial clinic visit and follow-up visit after completion of speech therapy. Typically a time scale of 6-12 weeks depending on how soon speech/swallow/upper airway therapy is started.
  The Vocal Handicap Index-10 (VHI-10) will be used to obtain a quick, reliable, and quantifiable measure of patients' own vocal handicap perception. In 2004, Rosen et al designed a new shortened version of the first and broadly used global handicap assessment tool for voice disorders, the VHI. This questionnaire comprises 10 questions from the original 30 questions of the VHI and was called the VHI-10. The VHI-10 is a powerful representation of the VHI (30 items) to quantify patients' perception of their voice handicap. The VHI-10 has also been shown to be reliable, valid, and sensitive in a wide range of voice disorders (Rosen et al., 2004). This has a minimum value of 0 and a maximum value of 40. A higher score means a worse outcome.
Change in Eating Assessment Tool-10 Score Following Therapy | Recorded at initial clinic visit and follow-up visit after completion of speech therapy. Typically a time scale of 6-12 weeks depending on how soon speech/swallow/upper airway therapy is started.
  The EAT-10 is a 10-question self-assessment tool to identify adults who exhibit signs and symptoms that may be indicative of dysphagia and who may require further referral. The EAT-10 has begun to be used in research with older adults in different settings, including an aged care facility (Wakabayashi & Matsushima, 2016), acute hospital care (Matsuo, Yoshimura, Ishizaki, & Ueno, 2016), and the community (Momoki et al., 2017). In the aged care setting, EAT-10 results suggesting the presence of dysphagia have been shown to be independently associated with a risk of malnutrition and impaired functional status (Wakabayashi & Matsushima, 2016). This has a minimum value of 0 and a maximum value of 40. A higher score means a worse outcome.
Change in Cough Severity Index Score Following Therapy | Recorded at initial clinic visit and follow-up visit after completion of speech therapy. Typically a time scale of 6-12 weeks depending on how soon speech/swallow/upper airway therapy is started.
  Cough Severity Index (CSI) is a short and self-administered questionnaire for patients with self-perceived symptoms of cough in order to quantify severity of chronic cough relating to upper airway disease and facilitate treatment outcomes. CSI helps quantify severity of cough in patients with chronic cough (CC) related to the upper airway. This has a minimum value of 0 and a maximum value of 40. A higher score means a worse outcome.
Change in Dyspnea Index Score Following Therapy | Recorded at initial clinic visit and follow-up visit after completion of speech therapy. Typically a time scale of 6-12 weeks depending on how soon speech/swallow/upper airway therapy is started.
  Dyspnea Index (DI) is intended to serve as a quick and efficient patient-completed questionnaire to measure upper-airway related symptoms. The DI, by traditional psychometric standards, has good psychometric properties for patients with symptoms of upper airway dyspnea. This has a minimum value of 0 and a maximum value of 40. A higher score means a worse outcome.

SECONDARY OUTCOMES:
Change in Voice Fundamental Frequency as Measured in the VoiceEvalu8 App Following Therapy | Recorded at initial clinic visit and follow-up visit after completion of speech therapy. Typically a time scale of 6-12 weeks depending on how soon speech/swallow/upper airway therapy is started.
  Candidates of voice and/or upper-airway therapy will be assessed by acoustic instruments that record and analyze the speaker's voice. Standard clinical measures will be taken.
Change in Voice Cepstral Peak Prominence (CPP) as Measured in the VoiceEvalu8 App Following Therapy | Recorded at initial clinic visit and follow-up visit after completion of speech therapy. Typically a time scale of 6-12 weeks depending on how soon speech/swallow/upper airway therapy is started.
  Candidates of voice and/or upper-airway therapy will be assessed by acoustic instruments that record and analyze the speaker's voice. Standard clinical measures will be taken.
Change in Acoustic Voice Quality Index (AVQI) as Measured in the VoiceEvalu8 App Following Therapy | Recorded at initial clinic visit and follow-up visit after completion of speech therapy. Typically a time scale of 6-12 weeks depending on how soon speech/swallow/upper airway therapy is started.
  Candidates of voice and/or upper-airway therapy will be assessed by acoustic instruments that record and analyze the speaker's voice. Standard clinical measures will be taken.
Change in Iowa Oral Performance Instrument (IOPI) Following Therapy | Recorded at initial clinic visit and follow-up visit after completion of speech therapy. Typically a time scale of 6-12 weeks depending on how soon speech/swallow/upper airway therapy is started.
  Candidates of swallowing therapy (patients with dysphagia) will undergo standard instrumental swallowing assessment to assess tongue strength.
Change in DIGEST Scale Score Following Therapy | Recorded at initial clinic visit and follow-up visit after completion of speech therapy. Typically a time scale of 6-12 weeks depending on how soon speech/swallow/upper airway therapy is started.
  Candidates of swallowing therapy (patients with dysphagia) will undergo standard instrumental swallowing assessment to assess tongue strength and swallowing safety. The minimum score is a 0 and the maximum score is a 4. A higher score is a worse outcome and poorer swallowing safety.
Change in Functional Oral Intake Scale (FOIS) Score Following Therapy | Recorded at initial clinic visit and follow-up visit after completion of speech therapy. Typically a time scale of 6-12 weeks depending on how soon speech/swallow/upper airway therapy is started.
  Candidates of swallowing therapy (patients with dysphagia) will undergo standard instrumental swallowing assessment to assess tongue strength and swallow function. The minimum score is a 1 and the maximum score is a 7. A 7 means a better outcome/diet without restrictions. A 1 would mean no intake orally.

CONTACTS AND LOCATIONS:
Overall Officials: Clark Rosen, MD, Principal Investigator — University of California, San Francisco
Locations (4):
- United States (4):
  - UCSF Voice and Swallowing Center, San Francisco, California
  - Emory Voice Center, Atlanta, Georgia
  - NYU Voice Center, New York, New York
  - Cornell Medical Center, New York, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Leclerc AA, Gillespie AI, Tadic SD, Smith LJ, Rosen CA. The prevalence of cognitive impairment in laryngology treatment-seeking patients. Laryngoscope. 2020 Aug;130(8):2003-2007. doi: 10.1002/lary.28355. Epub 2019 Oct 25. PMID 31654439
- [Background] Shembel AC, Rosen CA, Zullo TG, Gartner-Schmidt JL. Development and validation of the cough severity index: a severity index for chronic cough related to the upper airway. Laryngoscope. 2013 Aug;123(8):1931-6. doi: 10.1002/lary.23916. Epub 2013 Jun 4. PMID 23737389
- [Background] Gartner-Schmidt JL, Shembel AC, Zullo TG, Rosen CA. Development and validation of the Dyspnea Index (DI): a severity index for upper airway-related dyspnea. J Voice. 2014 Nov;28(6):775-82. doi: 10.1016/j.jvoice.2013.12.017. Epub 2014 Oct 12. PMID 25311596
- [Background] Gartner-Schmidt J, Rosen C. Treatment success for age-related vocal fold atrophy. Laryngoscope. 2011 Mar;121(3):585-9. doi: 10.1002/lary.21122. Epub 2010 Aug 3. PMID 21344441
- [Background] Misono S, Yueh B, Stockness AN, House ME, Marmor S. Minimal Important Difference in Voice Handicap Index-10. JAMA Otolaryngol Head Neck Surg. 2017 Nov 1;143(11):1098-1103. doi: 10.1001/jamaoto.2017.1621. PMID 28973078